CLINICAL TRIAL: NCT04039607
Title: A Randomized, Multi-center, Phase 3 Study of Nivolumab in Combination With Ipilimumab Compared to Sorafenib or Lenvatinib as First-Line Treatment in Participants With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Nivolumab in Combination With Ipilimumab in Participants With Advanced Hepatocellular Carcinoma
Acronym: CheckMate 9DW
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9DW
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Ipilimumab; Sorafenib; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Sorafenib/lenvatinib (Active Comparator)
  Interventions: Drug: Sorafenib; Drug: lenvatinib

INTERVENTIONS:
Drug: Nivolumab — Participants will receive nivolumab as intravenous (IV) infusion.
  Arms: Nivolumab + Ipilimumab
Drug: Ipilimumab — Participants will receive ipilimumab as IV infusion.
  Arms: Nivolumab + Ipilimumab
Drug: Sorafenib — Participants will receive sorafenib as oral tablets.
  Arms: Sorafenib/lenvatinib
Drug: lenvatinib — Participants will receive lenvatinib as oral capsules.
  Arms: Sorafenib/lenvatinib

SUMMARY:
The main purpose of this study is to compare the overall survival (OS) of nivolumab plus ipilimumab versus standard of care (SOC) (sorafenib or lenvatinib) in all randomized participants with advanced hepatocellular carcinoma (HCC) who have not received prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of HCC based on histological confirmation
* Participants must have an advanced HCC
* Participants must have at least one Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 measurable previously untreated lesion
* Child-Pugh score 5 or 6
* Eastern Cooperative Oncology Group (ECOG) performance status(PS) 0 or 1

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Prior liver transplant
* Episodes of hepatic encephalopathy (greater than or equal to [>=] Grade 2) within 12 months prior to randomization
* Active brain metastases or leptomeningeal metastases

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 4 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 4 years
Duration of Response (DOR) | Up to 4 years
Time to Symptom Deterioration (TTSD) | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (210):
- United States (15):
  - Local Institution - 0292, Tucson, Arizona
  - Local Institution - 0288, Coronado, California
  - Local Institution - 0157, Duarte, California
  - Local Institution - 0077, Washington D.C., District of Columbia
  - Local Institution - 0027, Louisville, Kentucky
  - Local Institution - 0190, Baltimore, Maryland
  - Local Institution, Ann Arbor, Michigan
  - Local Institution - 0018, Detroit, Michigan
  - Local Institution - 0295, Newark, New Jersey
  - Local Institution - 0043, Toledo, Ohio
  - Local Institution - 0284, Pittsburgh, Pennsylvania
  - Local Institution - 0304, Dallas, Texas
  - Local Institution - 0202, Houston, Texas
  - Local Institution - 0046, Lubbock, Texas
  - Local Institution - 0172, Salt Lake City, Utah
- Argentina (5):
  - Local Institution - 0037, Caba, Buenos Aires
  - Local Institution - 0194, Pilar, Buenos Aires
  - Local Institution - 0282, Rosario, Santa Fe Province
  - Local Institution - 0136, Buenos Aires
  - Local Institution - 0058, San Miguel de Tucumán
- Australia (10):
  - Local Institution - 0003, Kogarah, New South Wales
  - Local Institution - 0038, Liverpool, New South Wales
  - Local Institution - 0002, Westmead, New South Wales
  - Local Institution - 0004, Birtinya, Queensland
  - Local Institution - 0013, Herston, Queensland
  - Local Institution - 0009, Adelaide, South Australia
  - Local Institution - 0019, Clayton, Victoria
  - Local Institution - 0026, Fitzroy, Victoria
  - Local Institution - 0001, Melbourne, Victoria
  - Local Institution - 0020, St Albans, Victoria
- Austria (5):
  - Local Institution - 0114, Sankt Pölten, Lower Austria
  - Local Institution - 0057, Wiener Neustadt, Lower Austria
  - Local Institution - 0188, Graz
  - Local Institution - 0065, Klagenfurt
  - Local Institution - 0186, Vienna
- Belgium (7):
  - Local Institution - 0034, Brussels
  - Local Institution - 0008, Federal District
  - Local Institution - 0124, Ghent
  - Local Institution - 0298, Ghent
  - Local Institution - 0099, Haine-Saint-Paul
  - Local Institution - 0064, Leuven
  - Local Institution - 0104, Liège
- Brazil (13):
  - Local Institution - 0278, Vitória, Espírito Santo
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution - 0061, Salvador, Estado de Bahia
  - Local Institution - 0181, Brasília, Federal District
  - Local Institution - 0279, Ijuí, Rio Grande do Sul
  - Local Institution - 0060, Pelotas, Rio Grande do Sul
  - Local Institution - 0054, Jaú, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Local Institution - 0016, Paranã
  - Local Institution - 0015, Rio de Janeiro
  - Local Institution - 0023, São Paulo
  - Local Institution - 0022, São Paulo
  - Local Institution - 0050, São Paulo
- Local Institution - 0192, Edmonton, Alberta, Canada
- Chile (8):
  - Local Institution - 0094, La Serena, Coquimbo Region
  - Local Institution - 0296, Temuco, Región de la Araucanía
  - Local Institution - 0012, Viña del Mar, Región de Valparaíso
  - Local Institution - 0216, Viña del Mar, Región de Valparaíso
  - Local Institution - 0283, Santiago, RM
  - Local Institution - 0095, Santiago, Santiago Metropolitan
  - Local Institution - 0024, Santiago, Santiago Metropolitan
  - Local Institution - 0156, Santiago, Santiago Metropolitan
- China (27):
  - Local Institution - 0120, Hefei, Anhui
  - Local Institution - 0146, Hefei, Anhui
  - Local Institution - 0175, Beijing, Beijing Municipality
  - Local Institution - 0152, Beijing, Beijing Municipality
  - Local Institution - 0151, Fuzhou, Fujian
  - Local Institution - 0121, Fuzhou, Fujian
  - Local Institution - 0125, Guangzhou, Guangdong
  - Local Institution - 0150, Guangzhou, Guangdong
  - Local Institution - 0135, Harbin, Heilongjiang
  - Local Institution - 0109, Changsha, Hunan
  - Local Institution - 0059, Changsha, Hunan
  - Local Institution - 0130, Nanjing, Jiangsu
  - Local Institution - 0145, Nanchang, Jiangxi
  - Local Institution - 0149, Nanchang, Jiangxi
  - Local Institution - 0162, Changchun, Jilin
  - Local Institution - 0166, Changchun, Jilin
  - Local Institution - 0131, Dalian, Liaoning
  - Local Institution - 0123, Shenyang, Liaoning
  - Local Institution - 0132, Shenyang, Liaoning
  - Local Institution - 0133, Xi'an, Shaanxi
  - Local Institution - 0147, Xi'an, Shan3xi
  - Local Institution - 0307, Xi'an, Shan3xi
  - Local Institution - 0153, Qingdao, Shandong
  - Local Institution - 0134, Shanghai, Shanghai Municipality
  - Local Institution - 0179, Chongqing, Sichuan
  - Local Institution - 0108, Hangzhou, Zhejiang
  - Local Institution - 0107, Hangzhou, Zhejiang
- Czechia (2):
  - Local Institution - 0274, Prague, Prague
  - Local Institution, Brno
- France (14):
  - Local Institution - 0068, Amiens
  - Local Institution - 0116, Caen
  - Local Institution - 0069, Clichy
  - Local Institution - 0138, Dijon
  - Local Institution - 0081, Grenoble
  - Local Institution - 0070, Lyon
  - Local Institution, Marseille
  - Local Institution - 0082, Montpellier
  - Local Institution - 0067, Nice
  - Local Institution - 0025, Pessac
  - Local Institution - 0137, Poitiers
  - Local Institution - 0042, Toulouse
  - Local Institution - 0071, Vandœuvre-lès-Nancy
  - Local Institution - 0051, Villejuif
- Germany (12):
  - Local Institution - 0005, Frankfurt am Main, Hesse
  - Local Institution - 0231, Bonn
  - Local Institution - 0028, Cologne
  - Local Institution - 0052, Essen
  - Local Institution - 0185, Freiburg im Breisgau
  - Local Institution - 0006, Hamburg
  - Local Institution - 0102, Hanover
  - Local Institution - 0118, Leipzig
  - Local Institution - 0031, Mainz
  - Local Institution - 0056, Mannheim
  - Local Institution, München
  - Local Institution - 0053, North Rhine-Westphalia
- Hong Kong (2):
  - Local Institution - 0036, Hong Kong
  - Local Institution - 0032, Hong Kong
- Italy (11):
  - Local Institution - 0110, Meldola, Forli-Cesena
  - Local Institution - 0101, Rozzano, Milano
  - Local Institution - 0084, Candiolo
  - Local Institution - 0039, Milan
  - Local Institution - 0100, Novara
  - Local Institution - 0219, Padua
  - Local Institution - 0033, Parma
  - Local Institution - 0112, Roma
  - Local Institution - 0079, Rome
  - Local Institution - 0111, Siena
  - Local Institution - 0044, Vicenza
- Japan (20):
  - Local Institution - 0193, Kashiwa-shi, Chiba
  - Local Institution - 0203, Matsuyama, Ehime
  - Local Institution - 0176, Kanazawa, Ishikawa-ken
  - Local Institution - 0200, Yokohama, Kanagawa
  - Local Institution - 0262, Yokohama, Kanagawa
  - Local Institution - 0189, Kyoto, Kyoto
  - Local Institution - 0261, Kashihara, Nara
  - Local Institution - 0263, Abeno-ku, Osaka
  - Local Institution - 0127, Sayama, Osaka
  - Local Institution - 0281, Saga, Saga-ken
  - Local Institution - 0258, Iruma-gun, Saitama
  - Local Institution - 0259, Izunokuni-shi, Shizuoka
  - Local Institution - 0128, Minato, Tokyo
  - Local Institution - 0122, Minato-ku, Tokyo
  - Local Institution - 0201, Mitaka, Tokyo
  - Local Institution - 0199, Musashino-shi, Tokyo
  - Local Institution - 0204, Chiba
  - Local Institution - 0178, Fukuoka
  - Local Institution - 0177, Hiroshima
  - Local Institution - 0155, Sapporo
- New Zealand (2):
  - Local Institution - 0286, Christchurch, Canterbury
  - Local Institution - 0047, Auckland
- Poland (3):
  - Local Institution - 0148, Gdansk
  - Local Institution - 0049, Otwock
  - Local Institution - 0092, Warsaw
- Puerto Rico (2):
  - Local Institution - 0289, Rio Piedras
  - Local Institution - 0035, San Juan
- Romania (5):
  - Local Institution - 0103, Craiova, Dolj
  - Local Institution - 0164, Bucharest
  - Local Institution - 0165, Cluj-Napoca
  - Local Institution, Craiova
  - Local Institution - 0163, Timișoara
- Russia (8):
  - Local Institution - 0029, Arkhangelsk
  - Local Institution - 0066, Barnaul
  - Local Institution - 0074, Chelyabinsk
  - Local Institution - 0007, Moscow
  - Local Institution - 0072, Pyatigorsk
  - Local Institution - 0075, Saint Petersburg
  - Local Institution - 0091, Saint Petersburg
  - Local Institution - 0073, Sochi
- Singapore (3):
  - Local Institution - 0048, Singapore
  - Local Institution - 0017, Singapore
  - Local Institution - 0174, Singapore
- South Korea (9):
  - Local Institution - 0143, Seongnam-si, Gyeonggi-do
  - Local Institution - 0167, Guro-gu, Seoul
  - Local Institution - 0062, Jongno-gu, Seoul
  - Local Institution - 0142, Busan
  - Local Institution - 0097, Gyeonggi-do
  - Local Institution - 0098, Gyeongsangnam-do
  - Local Institution - 0141, Seoul
  - Local Institution - 0140, Seoul
  - Local Institution - 0139, Seoul
- Spain (12):
  - Local Institution - 0297, Barcelona
  - Local Institution - 0055, Barcelona
  - Local Institution - 0089, Barcelona
  - Local Institution - 0090, Córdoba
  - Local Institution - 0087, El Palmar
  - Local Institution - 0041, Madrid
  - Local Institution - 0093, Madrid
  - Local Institution - 0290, Madrid
  - Local Institution - 0045, Majadahonda
  - Local Institution - 0085, Pamplona
  - Local Institution - 0088, Santander
  - Local Institution - 0040, Zaragoza
- Local Institution - 0063, Bern, Switzerland
- Taiwan (9):
  - Local Institution - 0272, Kaohsiung City
  - Local Institution - 0096, Kaohsiung City
  - Local Institution - 0105, Taichung
  - Local Institution - 0271, Taichung
  - Local Institution - 0168, Tainan
  - Local Institution - 0270, Tainan
  - Local Institution - 0144, Taipei
  - Local Institution - 0078, Taipei
  - Local Institution - 0173, Taoyuan District
- United Kingdom (4):
  - Local Institution - 0171, London, Greater London
  - Local Institution - 0154, Guildford, Surrey
  - Local Institution - 0160, Edinburgh
  - Local Institution - 0129, London

REFERENCES:
- [Derived] Yau T, Galle PR, Decaens T, Sangro B, Qin S, da Fonseca LG, Karachiwala H, Blanc JF, Park JW, Gane E, Pinter M, Pena AM, Ikeda M, Tai D, Santoro A, Pizarro G, Chiu CF, Schenker M, He A, Chon HJ, Wojcik-Tomaszewska J, Verset G, Wang QQ, Stromko C, Neely J, Singh P, Jimenez Exposito MJ, Kudo M; CheckMate 9DW investigators. Nivolumab plus ipilimumab versus lenvatinib or sorafenib as first-line treatment for unresectable hepatocellular carcinoma (CheckMate 9DW): an open-label, randomised, phase 3 trial. Lancet. 2025 May 24;405(10492):1851-1864. doi: 10.1016/S0140-6736(25)00403-9. Epub 2025 May 8. PMID 40349714
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04039607.html